CLINICAL TRIAL: NCT03137849
Title: Autonomic and Cardiovascular Changes of Yoga Poses, Breath Control and Stretching Exercises in Hypertensive Post-Menopause Women: Randomized Controlled Trial
Brief Title: Yoga Poses and Breath Control Cardiovascular Changes in Hypertensive Post-Menopause Women
Acronym: YOGINI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: 5273/16
Record Dates: First submitted 2017-03-15; First posted 2017-05-03 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2017-07

CONDITIONS: Hypertension; Postmenopausal Symptoms
Keywords: Yoga; Hypertension; Post-Menopausal Women; Heart Rate Variability
MeSH Terms: conditions — Hypertension | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: All participants will be told they are attending to a yoga protocol. All outcomes assessments will be taken by blind investigators to the interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Yoga Poses + Breath control (Active Comparator): Twice a week 75 minutes video class of yoga poses routine ( including yoga bandhas with specific muscles contractions) combined with ujjayi pranayama technique as breath control
  Interventions: Other: Yoga Poses; Other: Breath Control
- Yoga Poses (Active Comparator): Twice a week 75 minutes video class of yoga poses routine ( including yoga bandhas/ specific muscles contractions)
  Interventions: Other: Yoga Poses
- Stretching Exercises + Breath control (Active Comparator): Twice a week 75 minutes video class of stretching exercises routine combined with ujjayi pranayama technique as breath control
  Interventions: Other: Breath Control; Other: Stretching exercises
- Stretching Exercises (Active Comparator): Twice a week 75 minutes video class of stretching exercises routine
  Interventions: Other: Stretching exercises

INTERVENTIONS:
Other: Yoga Poses — Yoga poses routine including specific muscles contractions known as bandhas (pelvic floor, core and throat/neck contraction) within each pose, which are advised to be done with steadiness and comfort.
  Arms: Yoga Poses; Yoga Poses + Breath control
Other: Breath Control — Ujjayi pranayama (Victorious breath) Inhalation and exhalation are both done through the nose. The "ocean sound" is created by moving the glottis as air passes in and out. As the throat passage is narrowed so, too, is the airway, the passage of air through which creates a "rushing" sound. The length and speed of the breath is controlled by the diaphragm, the Strengthening of which is, in part, the purpose of ujjayi. The inhalations and exhalations are equal in duration.
  Arms: Stretching Exercises + Breath control; Yoga Poses + Breath control
Other: Stretching exercises — Stretching exercises routine based on dynamic and static exercises excluding those similar to yoga poses. This routine works on great range of motion of all body joints and main muscles groups/ chains.
  Arms: Stretching Exercises; Stretching Exercises + Breath control

SUMMARY:
Autonomic and endothelial imbalance in post menopause women raise the need to manage cardiovascular risk. Yoga poses and breathing control present controversial results on prevention and treatment of hypertension.. The aim of this study is to compare the effect of 12 week intervention based on yoga poses and their muscle contractions known as bandhas (pelvic floor, core and throat/neck) and ujjayi pranayama (victorious breath) on autonomic modulation, endothelial function, arterial stiffness, aerobic capacity and cognitive function of hypertensive post-menopausal women.

DETAILED DESCRIPTION:
Abstract: Increased hypertension prevalence in post-menopausal women, along with cardiovascular damages such as autonomic and endothelial imbalance raise the need to include non-pharmacological interventions, such as yoga in the management of cardiovascular risk. Yoga practices are composed by several variations of techniques including physical postures (yoga poses and specific muscles contractions), breathing control (pranayamas), relaxation and meditation, beside others.The effects of each of these compounds has not been elucidated up to date and can be considered confounding effects for commonly named "yoga programs". Existing yoga based data are controversial about its effect on prevention and treatment of hypertension and point to poor methodological standards of most studies. Considering the effects of comparable interventions such as slow breathing on improving autonomic modulation, resistive and isometric exercise on endothelial function, and associations of flexibility with arterial stiffness, it´s licit to search for specific effects of yoga compounds. Thus, the aim of this study is to compare the effect of 12 week intervention based on yoga poses including their muscle contractions known as bandhas (pelvic floor, core and throat/neck), ujjayi pranayama (victorious breath) and stretching/ flexibility on autonomic modulation, endothelial function, arterial stiffness, aerobic capacity and cognitive function of hypertensive post-menopausal women.

ELIGIBILITY:
Inclusion Criteria:

* FSH>35mui/ml
* minimum 12 months amenorrhea
* sedentary life style (less than 150 minutes per week of exercise)
* never been in yoga -practicing (self declaration)
* Blood pressure > 140/90 or in continuous use of medication (diuretics,Ca+ channel inhibitors, ACE inhibitors)

Exclusion Criteria:

* Use of Betablockers
* recent cardiovascular events or surgery
* renal alterations
* respiratory and/or motor pathologies
* smoking
* BMI>34,9

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-12-20 (Actual)

PRIMARY OUTCOMES:
Cardiovascular autonomic control by heart rate variability(HRV) and blood pressure variability (BPV) in frequency domain acquired by Finometer | 30 minutes
  Sympathovagal balance HRV (ratio of low frequency (LF in ms2) and high frequency (HF in ms2) components of HRV = LF/HF)

SECONDARY OUTCOMES:
Carotid -femoral pulse wave velocity (Complior) | 10 minutes
  Reduction of carotid -femoral pulse wave velocity (m/s)
Maximal Oxygen Uptake by Cardiopulmonary Exercise Test | 45 minutes
  Increase Maximal Oxygen Uptake (VO2max ml/kg/min)
Ambulatory Arterial Pressure Monitoring | 24 hours
  Decrease Ambulatory Arterial Pressure Monitoring (mmHg)
Respiratory rate and movements of rib cage and abdomen by Pneumotrace respiratory belt | 30 minutes along with Finometer
  Reduction of respiratory rate (cycles per minute/ cpm)
Blood samples laboratorial analysis | 5 minutes
  Improved blood sample analysis HDL cholesterol, glucose, creatinine, c-reactive protein (mg/dL)
Flow mediated dilation (FMD) of brachial artery by ultrasound | 20 minutes
  Increase Flow Mediated Dilation (FMD) (%)
Fat percentage by Bioimpedance | 5 minutes
  Reduction of fat percentage and increase of lean mass (% )
Cognitive function | 40 minutes
  Changes in scores of Mini Mental State Examination (0 to 30)
Diaphragm Thickness by ultrasound | 5 minutes
  Increase diaphragm thickness (mm)
Intima Media Thickness of carotid artery by ultrasound | 5 minutes
  Decrease of intima media thickness (IMT) (mm)
Blood sample analysis of oxidative stress markers (Spectrophotometry) | 5 minutes along for all blood samples
  Levels of Superoxide Dismutase (SOD) (un/SOD/mg protein)
Blood levels of sample analysis of Inflammatory markers (ELISA) | 5 minutes along for all blood samples
  Levels of Interleukin(IL) IL 1, IL 6, IL 10 (pg/ml)Tumor Necrosis Factor (TNF) alpha (pg/ml)
Assessment of center of pressure (COP) and balance by baropodometry platform | 5 minutes
  Decreased area of COP (cm2)
Sit and reach flexibility test | 5 minutes
  Increase flexibility levels (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cláudia Irigoyen, PhD, Study Director — Institute of Cardiology/ University Foundation of Cardiology
Locations (1):
- Cardiology Institute of Rio Grande do Sul, Pôrto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided